CLINICAL TRIAL: NCT04795115
Title: Feasibility and Acceptability of an Auditory Rhythmical Cueing Intervention Targeting Balance and Gait in Early Rehabilitation (ARCAS)
Brief Title: The ARCAS Study: Auditory Rhythmical Cueing for Gait in Acute Stroke
Acronym: ARCAS
Status: Completed | Type: Observational
Sponsor: Northumbria Healthcare NHS Foundation Trust (Other)
Responsible Party: Sponsor
Other Study IDs: 0031
Record Dates: First submitted 2019-01-09; First posted 2021-03-12 (Actual); Last update posted 2021-03-12 (Actual); Status verified 2021-03

CONDITIONS: Stroke
MeSH Terms: conditions — Stroke

STUDY DESIGN:
Observational Model: Other | Time Perspective: Other
Patient Registry: Yes
Target Follow-Up Duration: 3 Weeks
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

INTERVENTIONS:
Other: Auditory rhythmical cueing — Auditory rhythmical cueing intervention targeting balance and gait for 30 minutes x5 per week for 3 weeks.

SUMMARY:
Difficulties with walking is a common and distressing problem following stroke and can lead to reduced independence. Research suggests that using an auditory cue, such as a regular beat or pulse, as part of rehabilitation can improve walking. It is also recommended that early rehabilitation following stroke delivers the bestoutcome for patients.

Study aim:To determine whether the use of auditory cueing in early stroke rehabilitation is feasible during a balance and gait therapy programme.

Study participants: Adults following acute stroke with walking problems. Participants must be able to sit unsupported and stand with assistance of 1 or 2 people. They will be recruited from the acute stroke unit at North Tyneside General Hospital 2 days to 4 weeks following stroke. A total of 12 participants will be recruited.

Study setting: Acute stroke unit - North Tyneside General Hospital and participants homes if they are discharged within the study period.

Intervention:Participants will receive auditory rhythmical cueing intervention targeting balance and gait for 30 minutes x5 / week for 3 weeks within the physiotherapy gym on the stroke unit or at home if discharged within the intervention period. The 30 minutes will consist of balance exercises and walking practice using auditory cueing with a metronome.

Measures:1. What the participants and the therapists think of the intervention will be assessed by questionnaires. The questionnaires contain open and closed questions and have been developed specifically for this study.

2.The stroke survivors trunk control, balance and walking will be assessed before and after the intervention.

Study Duration: 12 months

Future Plans: This study will be used to inform a larger study testing if the intervention works and how much it costs

ELIGIBILITY:
Inclusion Criteria:

* Adults (> 18 years) following acute stroke (any subtype) with residual mobility problems
* Within 2 days - 4 weeks post-stroke.
* Be able to sit unsupported and stand with assistance of 1 or 2 people
* Able to provide informed consent to participate in the study.

Exclusion Criteria:

* Unable to follow the intervention due to cognitive or language impairment.
* Other medical problems affecting walking and balance (e.g. Parkinson's Disease, severe osteoarthritis and cardiopulmonary conditions).

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Adults within 2 days to 3 weeks following acute stroke with residual mobility problems. They must be able to sit unsupported, stand with assistance of 1- 2 people and be able to comply with the intervention programme.
Sampling Method: Non-Probability Sample
Enrollment: 12 (Actual)
Dates: Start 2019-02-04 (Actual); Primary Completion 2019-05-31 (Actual); Study Completion 2019-08-08 (Actual)

PRIMARY OUTCOMES:
Participant questionnaire | 3 weeks
  To seek views of patients on the intervention programme
Therapist questionnaire | 3 weeks
  To seek views from therapists on the intervention programme

OTHER OUTCOMES:
Functional Ambulatory category | 3 weeks
  Functional walking test that evaluates ambulation ability - score 0-5
Trunk Impairment Scale | 3 weeks
  measures trunk control - Score 0-23
Trunk ControlTest | 3 weeks
  To assess motor impairment - Score 0-100

CONTACTS AND LOCATIONS:
Locations (1):
- North Tyneside General Hospital, Newcastle upon Tyne, Tyne and Wear, United Kingdom

IPD SHARING:
Plan to Share IPD: Undecided